CLINICAL TRIAL: NCT03492086
Title: Clinical Study to Evaluate the Effectiveness and Safety of the Consumption of a Food Supplement in a Group of Healthy People
Brief Title: Study of the Consumption of a Food Supplement in a Group of Healthy People
Acronym: FORCANCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMD PI0017
Record Dates: First submitted 2018-03-19; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Immune System and Related Disorders
Keywords: Rosmarinus officinalis L; alkylglycerols; immuno-nutrition; colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosemary and alkylglycerol capsules (Experimental)
  Interventions: Dietary Supplement: Dietary supplementation with capsules containing rosemary and alkylglycerol
- Control capsules (Placebo Comparator)
  Interventions: Dietary Supplement: Dietary supplementation with control capsules

INTERVENTIONS:
Dietary Supplement: Dietary supplementation with capsules containing rosemary and alkylglycerol
  Arms: Rosemary and alkylglycerol capsules
Dietary Supplement: Dietary supplementation with control capsules
  Arms: Control capsules

SUMMARY:
Bioactive supplements might display relevant therapeutic properties according to validated molecular effects. Herein, the effect of a supplement based on diterpenes from Rosmarinus Officinalis L. and alkylglycerols with proven properties against signaling pathways involved in tumorigenesis is evaluated. The biological and molecular effects of this supplement, mainly based on expected effects on immune and genetic modulatory properties is investigated. For this purpose, 60 healthy volunteers were enrolled in a six week, double-blind, randomized and parallel pilot study with two study arms -rosemary and alkylglycerol containing capsules and control capsules. The study includes the analysis of (1) immunological parameters (ex vivo cytokine profile of LPS stimulated PBMC and PBMC phenotyping by cluster differentiation (CD) markers), (2) regulation of the expression of genes linked to immuno-modulation, inflammation, oxidative stress response and cancer, and (3) the analysis of correlation of selected genetic variants (SNPs) with the differential responses among individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years
* Adequate understanding of the study.
* Willingness to complete the entire treatment.

Exclusion Criteria:

* BMI >30
* Diagnosis of type 2 diabetes mellitus (T2D), hypertension, dyslipidemia or other cardiometabolic disorders
* Impaired cognitive function;
* Diagnosed hepatic, renal, or cardiovascular disease
* Subjects with primary immunodeficiency disorders, consumption of drugs with influence on the immune system, splenectomy.
* Presence of other pathologies like asthma, food allergies, Crohn's, myasthenia gravis, lupus
* Consumption of vitamins, minerals, supplements of antioxidant extracts or protein supplements in the 2 weeks prior to the start of the study
* Subjects treated with drugs affecting the lipid or glycemic profile during the previous 30 days
* Consumption of anticoagulants or antiplatelet agents, cyclosporine, acetylsalicylic acid, antihistamines or sedatives
* Hypersensitivity to rosemary, to its components or other members of the family of lipped plants or to soybean as excipient of the capsules
* Allergy or hypersensitivity to fish
* Habitual smoking or high consumption alcohol
* Pregnant or lactating women
* High-intensity physical exercise.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2015-12-22 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
Changes in ex vivo cytokine profile produced by lipopolysaccharide (LPS)-stimulated peripheral blood mononuclear cells (PBMCs) | Baseline and after 6 weeks of treatment
  Isolated PBMCs were first incubated for 12h, and then after LPS treated. Supernatants were recovered to determine concentrations of Interleukin (IL) -1B, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IFNy and TNFa using a magnetic bead-based immunoassay (Human High Sensitivity T Cell Magnetic Bead Panel A MAGPIX-Luminex) kit from Millipore, following the manufacturer's instructions. A minimum of 50 beads per parameter was analyzed by the MAGPIX-Luminex system. Raw data (median ﬂuorescence intensity, MFI) were analyzed with the xPONENT software 4.1.

SECONDARY OUTCOMES:
Changes in oxidative stress status | Baseline and after 6 weeks
  To evaluate the changes in the oxidative stress the following biomarkers were measured in urine samples:
  * Oxidized-low density lipoproteins measured by sandwich enzyme-linked immunosorbent assay (ELISA) by using the monoclonal antibody mAb-4E6 (Mercodia AB, Sweden)
  * Isoprostanes and thromboxane B2 quantified by competitive ELISA (Enzo Biochem, Inc., NY, USA and Oxford Biomedical Research, MI, USA, respectively).
Changes in lipid profile | Baseline and after 6 weeks
  To evaluate lipid improvements the following measurements were considered: Triacylglycerol, Total Cholesterol, low Density Lipoprotein and High-Density Lipoprotein measured by routine laboratory (CQS, Madrid, Spain, which follows the UNE-ISO 15189:2007 directives) methods.
Gene expression analysis | Baseline and after 6 weeks
  Gene-expression assays were performed in a HT-7900 Fast Real time PCR. GAPDH was used as endogenous control. RT-StatMiner software (Integromics® Inc., Madison, USA) was used to detect and determine the quality control and differential expression analyses. The Expression Suite Software (Life Technologies) program was used to obtain the Ct data. The ΔCt (Ct gene-CtGAPDH) was calculated and then the relative expression (RQ) between visits was calculated (V3-V1) following the 2-ΔΔCt method (Livak and Schmittgen 2001)
DNA genotyping | Baseline
  Genotyping was performed using the QuantStudio 12 K Flex Real-Time PCR System (Life Technologies Inc., Carlsbad, CA) with a TaqMan OpenArray plates. Single nucleotide polymorphisms (SNPs) involved in different parts of the pathogenic processes of inflammation, immune system, obesity, lipid metabolism, redox homeostasis and cancer, were analyzed using TaqMan Genotyper software.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Reglero, Proffesor, Study Director — IMDEA Food and Institute of Food Science Research (CIAL); Ana Ramirez de Molina, PhD, Principal Investigator — IMDEA Food
Locations (1):
- Viviana loria-Kohen, Madrid, Spain

REFERENCES:
- [Background] Al-Darmaki S, Knightshead K, Ishihara Y, Best A, Schenkein HA, Tew JG, Barbour SE. Delineation of the role of platelet-activating factor in the immunoglobulin G2 antibody response. Clin Diagn Lab Immunol. 2004 Jul;11(4):720-8. doi: 10.1128/CDLI.11.4.720-728.2004. PMID 15242947
- [Background] Deniau AL, Mosset P, Pedrono F, Mitre R, Le Bot D, Legrand AB. Multiple beneficial health effects of natural alkylglycerols from shark liver oil. Mar Drugs. 2010 Jul 19;8(7):2175-84. doi: 10.3390/md8072175. PMID 20714431
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Background] August DA, Huhmann MB; American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.) Board of Directors. A.S.P.E.N. clinical guidelines: nutrition support therapy during adult anticancer treatment and in hematopoietic cell transplantation. JPEN J Parenter Enteral Nutr. 2009 Sep-Oct;33(5):472-500. doi: 10.1177/0148607109341804. No abstract available. PMID 19713551
- [Background] Gonzalez-Vallinas M, Molina S, Vicente G, de la Cueva A, Vargas T, Santoyo S, Garcia-Risco MR, Fornari T, Reglero G, Ramirez de Molina A. Antitumor effect of 5-fluorouracil is enhanced by rosemary extract in both drug sensitive and resistant colon cancer cells. Pharmacol Res. 2013 Jun;72:61-8. doi: 10.1016/j.phrs.2013.03.010. Epub 2013 Apr 1. PMID 23557932
- [Background] Livak KJ, Schmittgen TD. Analysis of relative gene expression data using real-time quantitative PCR and the 2(-Delta Delta C(T)) Method. Methods. 2001 Dec;25(4):402-8. doi: 10.1006/meth.2001.1262. PMID 11846609
- [Background] Suchner U, Kuhn KS, Furst P. The scientific basis of immunonutrition. Proc Nutr Soc. 2000 Nov;59(4):553-63. doi: 10.1017/s0029665100000793. PMID 11115790